CLINICAL TRIAL: NCT01082913
Title: Study of the Effect of Sacral Surface Electrical Stimulation for Assisted Reproductive Technology
Brief Title: The Effect of Sacral Surface Electrical Stimulation for Assisted Reproductive Technology
Acronym: SSE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiga University (Other)
Responsible Party: Yoshihiko Shimizu, Shiga University of Medical Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSE
Record Dates: First submitted 2010-02-11; First posted 2010-03-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sacral Surface Electrical (SSE) (Experimental)
  Interventions: Device: SSE
- control (No Intervention)

INTERVENTIONS:
Device: SSE — Use of SSE or not use of SSE
  Arms: Sacral Surface Electrical (SSE)

SUMMARY:
The purpose of this study is to determine whether sacral surface electrical stimulation is effective in the treatment of assisted reproductive technology.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of infertility

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
thickness of myometrium after embryo transfer | 3 years

SECONDARY OUTCOMES:
implantation rate | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shiga University of Medical Science, Ohtsu, Shiga, Japan